CLINICAL TRIAL: NCT00085865
Title: PET Evaluation of Serotonin Transporters Using [C-11] DASB in Alcoholism
Brief Title: Serotonin Transporters in Alcoholism
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040208; 04-M-0208
Record Dates: First submitted 2004-06-15; First posted 2004-06-16 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-07

CONDITIONS: Alcoholism
Keywords: 5 HT; Neuroreceptors; Radiotracer; Neuroimaging; Serotonin Transporter; Alcoholism; PET; Healthy Volunteer; HV
MeSH Terms: conditions — Alcoholism

SUMMARY:
This study will compare serotonin transporter proteins in people with alcoholism and healthy volunteers to examine how these proteins may be related to the inability of people with alcoholism to appropriately regulate their alcohol consumption. Serotonin transporters regulate levels of the brain chemical serotonin. Problems in this regulation have been implicated in alcoholism.

Healthy normal volunteers and people who suffer from alcoholism who are between 18 and 75 years of age may be eligible for this study. Candidates are screened with a medical history and physical examination, psychiatric diagnostic interview, blood and urine tests, an electrocardiogram, urine toxicology screen, and written psychological evaluations.

Participants undergo positron emission tomography (PET) and magnetic resonance imaging (MRI) scanning to measure serotonin transporter levels in the brain.

PET uses small amounts of a radioactive chemical called a tracer that "labels" the serotonin transporters in the brain. The tracer used in this study is [11C]DASB. For the procedure, the subject lies on the scanner bed. A special mask is fitted to the head and attached to the bed to help keep the subject's head still during the scan so the images will be clear. A brief scan is done just before the radioactive tracer is injected. This scan provides measures of the brain that will help in the precise calculation of information from subsequent scans. After the tracer is injected through a catheter (plastic tube) placed in the arm, pictures are taken for about 2 hours.

MRI uses a magnetic field and radio waves to produce pictures of brain structure. The subject lies on a bed that slides into the tube-like scanner, wearing earplugs to muffle loud noises the machine makes when the magnetic fields are switched. The scan takes about an hour, during which time the subject can communicate with the technician.

DETAILED DESCRIPTION:
Alcoholism is characterized by the inability of individuals to regulate their consumption of alcohol appropriately. Serotonergic dysfunction has been implicated in the pathophysiology of this illness. Serotonin transporters (SERT) critically regulate the tone of serotonergic transmission (Gobbi et al 2001). In a brain imaging study using the SPECT radioligand, [123I] Beta-CIT, male alcoholics who had abstained from alcohol for more than four weeks, had significantly reduced serotonin transporters in the raphe area of the brainstem compared to healthy control subjects (Heinz et al 1998). However, the [123I] Beta-CIT ligand, binds with high affinity to both the dopamine transporter (DAT) and SERT. Binding of [123I] Beta-CIT in regions rich in SERT or DAT have been attributed to SERT and DAT respectively but in regions of mixed innervation (e.g. cortical regions), it is not possible to distinguish between SERT and DAT.

[11C]DASB is a PET ligand with high affinity for SERT with almost 1,000 fold selectivity versus DAT. Using this tracer, we will be able to measure SERT binding in cortical and subcortical brain regions including those with mixed innervation. [11C] DASB PET studies in humans (Houle et al 2000; Meyer et al 2001) indicate the feasibility of quantifying SERT binding in SERT rich regions. In the current protocol, we plan to use PET imaging with the radioligand, [11C] DASB, for serotonin transporter (SERT) to delineate regional abnormalities in SERT binding in two subject groups consisting of 30 patients with alcoholism and 30 healthy volunteers. Our goal of the present study is to further our understanding of the roles of the serotonergic systems in the pathophysiology of alcoholism.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Alcoholic and healthy subjects will be recruited from those screened by Dr. Daniel Hommer using either protocol (Protocol number 98-AA-0009) which is used to identify and recruit adult participants who meet DSM-IV criteria for alcohol dependence, alcohol abuse and healthy controls or protocol (Protocol number 05-AA-0121) assessment and treatment of people with alcohol drinking problems.

As stated in protocol 98-AA-0009, subjects will be recruited primarily from the Washington, DC metropolitan area through newspaper advertisements. These have been approved by the NIAAA IRB in the past and have not changed. As necessary these advertisements which are now primarily published in the Washington Post Health Section, will be reviewed and revised. Any revisions will be presented to the IRB. Subjects will also be recruited through outreach to health care professionals and treatment facilities throughout Northern Virginia, West Virginia and the Washington, DC and Baltimore metropolitan areas. Patient referrals for sources throughout the U.S. and on occasion international referrals also will be used.

Increased efforts will be made to recruit alcoholic subjects from the Hispanic community. This will take the form of contacts with treatment programs that serve Hispanic populations, as well as through advertising in Spanish language newspapers. We have decided to exclude children from this protocol because the NIH Clinical Center currently does not have any inpatient units capable of treating substance abusing patients who are under the age of 18. Every effort will be made to recruit a similar number of age-matched males and females. The two groups will not be individually matched by age. For example, we will not seek a control subject to match a particular alcoholic patient's age. Instead the two groups will be matched for mean age. We will obtain informed consent from all subjects per NIH guidelines for research studies.

INCLUSION CRITERIA - PATIENTS:

Age: 18-75

DSM-IV criteria for alcohol dependence or alcohol abuse.

INCLUSION CRITERIA - CONTROLS:

Age: 18-75

EXCLUSION CRITERIA:

PATIENTS AND CONTROLS:

Other current DSM-IV Axis I diagnostic criteria than alcohol dependence or alcohol abuse.

Psychotropic medication or other drugs that may cross the blood brain barrier.

Serious organic disease e.g. liver disease.

Claustrophobia.

Pregnancy.

Prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits.

Any condition that increases risk for MRI (e.g., pacemaker, metallic foreign body in the eye, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-06; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fujita M, Charney DS, Innis RB. Imaging serotonergic neurotransmission in depression: hippocampal pathophysiology may mirror global brain alterations. Biol Psychiatry. 2000 Oct 15;48(8):801-12. doi: 10.1016/s0006-3223(00)00960-4. PMID 11063976